CLINICAL TRIAL: NCT01529268
Title: Cysteamine Bitartrate Delayed-Release for the Treatment of Nonalcoholic Fatty Liver Disease (NAFLD) in Children (CyNCh)
Brief Title: Cysteamine Bitartrate Delayed-Release for the Treatment of NAFLD in Children
Acronym: CyNCh
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Cancer Institute (NCI) (NIH); Raptor Pharmaceuticals (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NASH-CyNCh; U01DK061718 (NIH); U01DK061728 (NIH); U01DK061731 (NIH); U01DK061732 (NIH); U01DK061734 (NIH); U01DK061737 (NIH); U01DK061738 (NIH); U01DK061730 (NIH); U01DK061713 (NIH)
Record Dates: First submitted 2012-01-18; First posted 2012-02-08 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2017-08

CONDITIONS: Nonalcoholic Fatty Liver Disease (NAFLD)
Keywords: Nonalcoholic Fatty Liver Disease (NAFLD); Cysteamine bitartrate delayed release; Children
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DR cysteamine bitartrate capsule (Active Comparator): Active DR cysteamine bitartrate capsule
  Interventions: Drug: DR cysteamine bitartrate capsule
- DR cysteamine bitartrate placebo (Placebo Comparator): Placebo DR cysteamine bitartrate capsule
  Interventions: Other: DR cysteamine bitartrate placebo

INTERVENTIONS:
Drug: DR cysteamine bitartrate capsule — * 600 mg/day (four 75 mg capsules twice daily) for patients ≤ 65 kg at baseline
  * 750 mg/day (five 75 mg capsules twice daily) for patients >65 - 80 kg at baseline
  * 900 mg/day (six 75 mg capsules twice daily) for patients >80 kg at baseline
  Other Names: cysteamine bitartrate delayed-release
  Arms: DR cysteamine bitartrate capsule
Other: DR cysteamine bitartrate placebo — * 600 mg/day (four 75 mg capsules twice daily) for patients ≤ 65 kg at baseline
  * 750 mg/day (five 75 mg capsules twice daily) for patients >65 - 80 kg at baseline
  * 900 mg/day (six 75 mg capsules twice daily) for patients >80 kg at baseline
  Arms: DR cysteamine bitartrate placebo

SUMMARY:
CyNCh is a multi-center, placebo-controlled clinical trial of children ages 8 to 17 years with biopsy-confirmed moderate to severe nonalcoholic fatty liver disease (NAFLD). The primary objective is to evaluate whether 52 weeks of treatment with cysteamine bitartrate delayed-release capsules will result in improvement in liver disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Children age 8-17 years
* Liver biopsy obtained within 90 days of screening visit and not more than 120 days before randomization
* Clinical history consistent with nonalcoholic fatty liver disease (NAFLD)
* Definite NAFLD based upon liver histology
* No evidence of any other liver disease by clinical history or histological evaluation
* A histological severity of: NAFLD Activity Score (NAS) ≥ 4.
* Sexually active female participants of childbearing potential (i.e., not surgically sterile [defined as tubal ligation, hysterectomy, or bilateral oophorectomy]) must agree to utilize the same two acceptable forms of contraception from screening through completion of the study and to complete a serum pregnancy test at each study visit. The acceptable forms of contraception for this study include hormonal contraceptives (oral, implant, transdermal patch, or injection) at a stable dose for at least 3 months prior to screening, and barrier (condom with spermicide, diaphragm with spermicide). Sexual activity will be ascertained at each study visit for post-menarchal females and if sexually active, subject must verify use of the same 2 acceptable forms of contraception. For pre-pubescent children, a documented attestation of abstinence from their parent or guardian will be acceptable.
* Participants must be able to swallow DR Cysteamine tablets with the tablet intact
* Written informed consent from parent or legal guardian
* Written informed assent from the child

Exclusion Criteria:

* There will be no exclusion criteria based on race, ethnicity or gender.
* Participants with a current history of the following conditions or any other health issues that make it unsafe for them to participate in the opinion of the Investigators:

  * Inflammatory bowel disease (if currently active) or prior resection of small intestine
  * Heart disease (e.g., myocardial infarction, heart failure, unstable arrhythmias)
  * Seizure disorder
  * Active coagulopathy
  * Gastrointestinal ulcers/bleeding
  * Renal dysfunction with a creatinine clearance < 90 mL/min/m2
  * History of active malignant disease requiring chemotherapy within the past 12 months prior to randomization
  * History of significant alcohol intake (AUDIT questionnaire) or inability to quantify alcohol consumption
  * Chronic use (more than 2 consecutive weeks) of medications known to cause hepatic steatosis or steatohepatitis (systemic glucocorticoids, tetracycline, anabolic steroids, valproic acid, salicylates, tamoxifen) in the past year.
  * The use of other known hepatotoxins within 90 days of liver biopsy or within 120 days of randomization
  * Initiation of medications with the intent to treat NAFLD/NASH in the time period following liver biopsy and prior to randomization
  * History of total parenteral nutrition (TPN) use in year prior to screening
  * History of bariatric surgery or planning to undergo bariatric surgery during study duration
  * Clinically significant depression (patients hospitalized for suicidal ideations or suicide attempts within the past 12 months)
  * Any female nursing, planning a pregnancy, known or suspected to be pregnant, or who has a positive serum pregnancy screen.
* Non-compensated liver disease with any one of the following hematologic, biochemical, and serological criteria on entry into protocol:

  * Hemoglobin < 10 g/dL;
  * White blood cell (WBC) < 3,500 cells/mm3 of blood;
  * Neutrophil count < 1,500 cells/mm3 of blood;
  * Platelets < 130,000 cells/mm3 of blood;
  * Direct bilirubin > 1.0 mg/dL
  * Total bilirubin >3 mg/dL
  * Albumin < 3.2 g/dL
  * International normalized ratio (INR) > 1.4
* Poorly controlled diabetes mellitus (hemoglobin A1c (HbA1c) > 9%)
* Evidence of other chronic liver disease:

  * Biopsy consistent with histological evidence of autoimmune hepatitis
  * Serum hepatitis B surface antigen (HBsAg) positive.
  * Serum hepatitis C antibody (anti-HCV) positive.
  * Iron/total iron binding capacity (TIBC) ratio (transferrin saturation) > 45% with histological evidence of iron overload
  * Alpha-1-antitrypsin (A1AT) phenotype ZZ or SZ
  * Wilson's disease
* Children who are currently enrolled in a clinical trial or who received an investigational study drug within 180 days of screening or liver biopsy.
* Subjects who are not able or willing to comply with the protocol or have any other condition that would impede compliance or hinder completion of the study, in the opinion of the investigator.
* Failure to give informed consent

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 169 (Actual)
Dates: Start 2012-06; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (10):
- United States (10):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago (NWU), Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - St. Louis University, St Louis, Missouri
  - Columbia University, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
  - University of Washington, Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Public use database deposited with the NIDDK Central Repository
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Currently available
Access Criteria: Apply through the NIDDK Central Repository: https://www.niddkrepository.org/home/
URL: https://repository.niddk.nih.gov/studies/cynch/?query=cynch

REFERENCES:
- [Derived] Jain AK, Buchannan P, Yates KP, Belt P, Schwimmer JB, Rosenthal P, Murray KF, Molleston JP, Scheimann A, Xanthakos SA, Behling CA, Hertel P, Nilson J, Neuschwander-Tetri BA, Tonascia J, Vos MB; Nonalcoholic Steatohepatitis Clinical Research Network (NASH CRN). Nutrition assessment and MASH severity in children using the Healthy Eating Index. Hepatol Commun. 2023 Dec 7;7(12):e0320. doi: 10.1097/HC9.0000000000000320. eCollection 2023 Dec 1. PMID 38055641
- [Derived] Schwimmer JB, Lavine JE, Wilson LA, Neuschwander-Tetri BA, Xanthakos SA, Kohli R, Barlow SE, Vos MB, Karpen SJ, Molleston JP, Whitington PF, Rosenthal P, Jain AK, Murray KF, Brunt EM, Kleiner DE, Van Natta ML, Clark JM, Tonascia J, Doo E; NASH CRN. In Children With Nonalcoholic Fatty Liver Disease, Cysteamine Bitartrate Delayed Release Improves Liver Enzymes but Does Not Reduce Disease Activity Scores. Gastroenterology. 2016 Dec;151(6):1141-1154.e9. doi: 10.1053/j.gastro.2016.08.027. Epub 2016 Aug 26. PMID 27569726
- See also: Nonalcoholic Steatohepatitis Clinical Research Network Centers — http://jhuccs1.us/nash/open/centers/centers.htm
- See also: The National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) — http://www2.niddk.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 10 NASH CRN clinical centers from June 2012 to January 2014.
Groups:
- DR Cysteamine Bitartrate Capsule: Active DR cysteamine bitartrate capsule
  DR cysteamine bitartrate capsule: ◦ 600 mg/day (four 75 mg capsules twice daily) for patients ≤ 65 kg at baseline
  * 750 mg/day (five 75 mg capsules twice daily) for patients >65 - 80 kg at baseline
  * 900 mg/day (six 75 mg capsules twice daily) for patients >80 kg at baseline
- DR Cysteamine Bitartrate Placebo: Placebo DR cysteamine bitartrate capsule
  DR cysteamine bitartrate placebo: ◦ 600 mg/day (four 75 mg capsules twice daily) for patients ≤ 65 kg at baseline
  * 750 mg/day (five 75 mg capsules twice daily) for patients >65 - 80 kg at baseline
  * 900 mg/day (six 75 mg capsules twice daily) for patients >80 kg at baseline
Period: Overall Study
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Started | 88 | 81
Completed 52-week Biopsy | 71 | 75
Completed | 76 | 78
Not Completed | 12 | 3
Not completed — Lost to Follow-up | 9 | 3
Not completed — Moved | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo | Total
Number analyzed (Participants) | 88 | 81 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (2.9) | 13.6 (2.5) | 13.7 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 63 | 56 | 119
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian/Alaska Native | 5 | 6 | 11
  Asian | 0 | 2 | 2
  Black or African-American | 3 | 3 | 6
  White | 56 | 46 | 102
  More than one race | 3 | 1 | 4
  Refusal/not stated | 21 | 23 | 44
Region of Enrollment [Number; unit: participants]
  United States | 88 | 81 | 169
Alanine aminotransferase [Mean (Standard Deviation); unit: U/L] | 140 (118) | 103 (76) | 123 (101)
Aspartate aminotransferase [Mean (Standard Deviation); unit: U/L] | 82 (71) | 59 (38) | 71 (59)
Weight group [Number; unit: participants]
  Less than or equal to 65 kg | 24 | 23 | 47
  >65-80 kg | 14 | 10 | 24
  >80 kg | 50 | 48 | 98

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Nonalcoholic Fatty Liver Disease (NAFLD)
Description: Centrally scored and masked assessment of histologic improvement in Nonalcholic Fatty Liver Disease (NAFLD) between the baseline liver biopsy and follow-up biopsy after 52 weeks of treatment, where improvement is defined as: (1) decrease in the NAFLD Activity Score (NAS) of 2 or more and (2) no worsening of fibrosis.
Time Frame: 52 weeks
Population: Analysis based on intention to treat; patients with missing 52-week biopsy were imputed as lack of improvement.
Measure: Number; unit: participants
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 88 | 81
participants | 25 | 18
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Test type: Superiority — Relative risks and p-values were calculated with the Cochran-Mantel-Haenszel chi-square tests, stratified by clinic and weight group, for binary outcomes; p = 0.34, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.3, 95% CI 2-sided [0.8 to 2.1]

2. Secondary Outcome: Change in Nonalcoholic Fatty Liver Disease (NAFLD) Activity Score (NAS)
Description: Change from baseline in the NAFLD Activity Score (NAS), which is a composite score equal to the sum of the steatosis grade (0-3), lobular inflammation grade (0-3), and hepatocellular ballooning grade (0-2), from centralized pathologist scoring of liver biopsies. The overall scale of the NAS is 0-8, with higher scores indicating more severe disease. The outcome measure, change from baseline in NAFLD Activity Score (NAS), has a possible range from -8 to +8, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome. Components of the NAS are scored as follows: Steatosis grade 0=<5% steatosis, 1=5-33% steatosis, 2=34-66% steatosis, 3=>66% steatosis. Lobular inflammation grade=amount of lobular inflammation (combines mononuclear, fat granulomas, and polymorphonuclear (pmn) foci): 0=0, 1=<2 under 20x magnification, 2=2-4 under 20x magnification, 3=>4 under 20x magnification. Hepatocellular ballooning 0=none, 1=mild, 2=more than mild.
Time Frame: 52 weeks
Population: The smaller number of participants analyzed is due to missing 52-week biopsies (complete case analysis).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 71 | 75
units on a scale | -0.8 (1.8) | -0.8 (1.8)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Test type: Superiority — P-values and mean changes from baseline were calculated using ANCOVA, regressing change from baseline to 52 weeks on treatment group and baseline value of the outcome, for outcome scores; p = 0.90, ANCOVA; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.6 to 0.5]

3. Secondary Outcome: Steatosis: Patients With Improvement
Description: Improvement in steatosis defined as any decrease in steatosis grade comparing 52-week biopsy to baseline.
Time Frame: 52 weeks
Population: Analysis based on intention to treat; patients with missing 52-week biopsy were imputed as lack of improvement.
Measure: Number; unit: participants
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 88 | 81
participants | 26 | 33
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Steatosis: patients with improvement; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.15, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.7, 95% CI 2-sided [0.5 to 1.1]

4. Secondary Outcome: Steatosis: Change in Score
Description: Change from baseline in steatosis score. Steatosis score is based on central pathologist grading of liver biopsies: 0=<5% steatosis; 1=5-33% steatosis, 2=34-66% steatosis, 3=>66% steatosis. Change in steatosis score has a possible range of -3 to +3, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome (no improvement).
Time Frame: 52 weeks
Population: The smaller number of participants analyzed is due to missing 52-week biopsies (complete case analysis).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 71 | 75
units on a scale | -0.3 (0.9) | -0.4 (0.9)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Steatosis: change in score; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.59, ANCOVA; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.2 to 0.4]

5. Secondary Outcome: Lobular Inflammation: Patients With Improvement
Description: Improvement in lobular inflammation defined as any decrease in lobular inflammation grade comparing 52-week biopsy to baseline.
Time Frame: 52 weeks
Population: Analysis based on intention to treat; patients with missing 52-week biopsy were imputed as lack of improvement.
Measure: Number; unit: participants
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 88 | 81
participants | 32 | 17
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.03, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.8, 95% CI 2-sided [1.1 to 2.9]

6. Secondary Outcome: Lobular Inflammation: Change in Score
Description: Change from baseline in lobular inflammation score. The amount of lobular inflammation is based on central pathologist grading of liver biopsies, and combines mononuclear, fat granulomas, and polymorphonuclear (pmn) foci: 0=none; 1=<2 under 20x magnification, 2=2-4 under 20x magnification, 3=>4 under 20x magnification. Change in lobular inflammation score has a possible range of -3 to +3, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome (no improvement).
Time Frame: 52 weeks
Population: The smaller number of participants analyzed is due to missing 52-week biopsies (complete case analysis).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 71 | 75
units on a scale | -0.4 (0.8) | -0.1 (0.8)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.06, ANCOVA; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.4 to 0.0]

7. Secondary Outcome: Hepatocellular Ballooning: Patients With Improvement
Description: Improvement in hepatocellular ballooning defined as any decrease in hepatocellular ballooning score comparing 52-week biopsy to baseline.
Time Frame: 52 weeks
Population: Analysis based on intention to treat; patients with missing 52-week biopsy were imputed as lack of improvement.
Measure: Number; unit: participants
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 88 | 81
participants | 17 | 21
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.29, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.8, 95% CI 2-sided [0.4 to 1.3]

8. Secondary Outcome: Hepatocellular Ballooning: Change in Score
Description: Change from baseline in hepatocellular ballooning score. The amount of hepatocellular ballooning is based on central pathologist grading of liver biopsies: 0=none; 1=few ballooned hepatocytes, 2=many ballooned hepatocytes. Change in hepatocellular ballooning score has a possible range of -2 to +2, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome (no improvement).
Time Frame: 52 weeks
Population: The smaller number of participants analyzed is due to missing 52-week biopsies (complete case analysis).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 71 | 75
units on a scale | -0.1 (0.7) | -0.3 (0.8)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.15, ANCOVA; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.1 to 0.3]

9. Secondary Outcome: Portal Inflammation: Patients With Improvement
Description: Improvement in portal inflammation defined as any decrease in portal inflammation score comparing 52-week biopsy to baseline.
Time Frame: 52 weeks
Population: Analysis based on intention to treat; patients with missing 52-week biopsy were imputed as lack of improvement.
Measure: Number; unit: participants
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 88 | 81
participants | 18 | 14
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.57, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.2, 95% CI 2-sided [0.6 to 2.3]

10. Secondary Outcome: Portal Inflammation: Change in Score
Description: Change from baseline in portal inflammation score. The amount of portal inflammation is based on central pathologist grading of liver biopsies: 0=none; 1=mild, 2=more than mild. Change in portal inflammation score has a possible range of -2 to +2, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome (no improvement).
Time Frame: 52 weeks
Population: The smaller number of participants analyzed is due to missing 52-week biopsies (complete case analysis).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 71 | 75
units on a scale | -0.1 (0.6) | -0.1 (0.6)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.76, ANCOVA; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.2]

11. Secondary Outcome: Fibrosis: Patients With Improvement
Description: Improvement in fibrosis stage defined as any decrease in fibrosis stage comparing 52-week biopsy to baseline.
Time Frame: 52 weeks
Population: Analysis based on intention to treat; patients with missing 52-week biopsy were imputed as lack of improvement.
Measure: Number; unit: participants
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 88 | 81
participants | 25 | 23
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.98, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.0, 95% CI 2-sided [0.6 to 1.6]

12. Secondary Outcome: Fibrosis: Change in Stage
Description: Change from baseline in fibrosis stage. The amount of fibrosis is based on central pathologist grading of liver biopsies: 0=none; 1a=mild, zone 3 perisinusoidal, 1b=moderate, zone 3, perisinusoidal, 1c=portal/periportal only, 2=zone 3 and periportal, any combination, 3=bridging, 4=cirrhosis. Fibrosis stages 1a, 1b, 1c recoded as 1, so the possible range of values for fibrosis stage was 0-4. Change in fibrosis stage has a possible range of -4 to +4, with negative values indicating a better outcome (improvement) and positive values indicating a worse outcome (no improvement).
Time Frame: 52 weeks
Population: The smaller number of participants analyzed is due to missing 52-week biopsies (complete case analysis).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 71 | 75
units on a scale | -0.3 (0.9) | -0.1 (1.0)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.24, ANCOVA; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.4 to 0.1]

13. Secondary Outcome: Resolution of NASH
Description: Patients with a change from a histological diagnosis of definite NASH or indeterminate for NASH to not NASH at end of treatment
Time Frame: 52 weeks
Population: Analysis was limited to patients with a diagnosis of definite NASH at baseline.
Measure: Number; unit: participants
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 24 | 23
participants | 4 | 2
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.29, Cochran-Mantel-Haenszel; Stratified by clinic and weight group; Risk Ratio (RR) = 2.7, 95% CI 2-sided [0.4 to 18.3]

14. Secondary Outcome: Change in Serum Aminotransferase and Gamma-glutamyl Transpeptidase
Time Frame: 52 weeks
Population: The smaller number of participants analyzed is due to missing 52-week laboratory data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 75 | 77
U/L
  Alanine aminotransferase | -53 (88) | -8 (77)
  Aspartate aminotransferase | -31 (52) | -4 (36)
  Gamma-glutamyl transpeptidase | -10 (23) | -1 (16)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Adjusted difference in mean changes in serum alanine aminotransferase (ALT). The change in ALT is adjusted for the baseline ALT value; therefore, the adjusted difference in mean changes is not equal to the net change; Test type: Superiority — P-value and difference in mean changes from baseline were calculated using ANCOVA models, regressing change from baseline to 52 weeks in serum alanine aminotransferase on treatment group and baseline value of serum alanine aminotransferase; p = 0.02, ANCOVA; Adjusted for baseline serum alanine aminotransferase; Adjusted difference in mean changes = -24, 95% CI 2-sided [-44 to -4]
Statistical Analysis 2: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Adjusted difference in mean changes in serum aspartate aminotransferase (AST). The change in AST is adjusted for the baseline AST value; therefore, the adjusted difference in mean changes is not equal to the net change; Test type: Superiority — P-value and difference in mean changes from baseline were calculated using ANCOVA models, regressing changes from baseline to 52 weeks in serum aspartate aminotransferase on treatment group and baseline value of serum aspartate aminotransferase; p = 0.008, ANCOVA; Adjusted for baseline serum aspartate aminotransferase; Mean Difference (Net) = -15, 95% CI 2-sided [-26 to -4]
Statistical Analysis 3: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Adjusted difference in mean changes in serum gamma-glutamyl transpeptidase (GGT). The change in GGT is adjusted for the baseline GGTvalue; therefore, the adjusted difference in mean changes is not equal to the net change; Test type: Superiority — P-value and difference in mean changes from baseline were calculated using ANCOVA models, regressing changes from baseline to 52 weeks in gamma-glutamyl transpeptidase on treatment group and baseline value of gamma-glutamyl transpeptidase; p = 0.02, ANCOVA; Adjusted for baseline gamma-glutamyl transpeptidase; Mean Difference (Net) = -7, 95% CI 2-sided [-13 to -1]

15. Secondary Outcome: Change in Weight (kg)
Time Frame: 52 weeks
Population: Smaller number of patients analyzed due to missing 52-week weight measurement.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 75 | 77
kg | 6.3 (9.3) | 7.8 (6.6)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Adjusted difference in mean changes in weight (kg). The change in weight is adjusted for the baseline weight value; therefore, the adjusted difference in mean changes is not equal to the net change; Test type: Non-Inferiority or Equivalence — P-value and adjusted difference in mean changes from baseline were calculated using ANCOVA models, regressing changes from baseline to 52 weeks in weight (kg) on treatment group and baseline weight (kg); p = 0.25, ANCOVA; Adjusted for baseline weight (kg); Adjusted difference in mean changes = -1.5, 95% CI 2-sided [-4.1 to 1.1]

16. Secondary Outcome: Change in Body-mass Index
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 75 | 77
kg/m^2 | 0.8 (2.8) | 1.1 (2.2)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Adjusted difference in mean changes in body mass index (BMI). The change in BMI is adjusted for the baseline BMI value; therefore, the adjusted difference in mean changes is not equal to the net change; Test type: Superiority — P-values and differences in mean changes from baseline were calculated using ANCOVA models, regressing changes from baseline to 52 weeks on treatment group and baseline value of the outcome; p = 0.42, ANCOVA; Adjusted for baseline BMI (kg/m2); Adjusted difference in mean changes = -0.3, 95% CI 2-sided [-1.1 to 0.5]

17. Secondary Outcome: Change in Body-mass Index Z-score
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: SD
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 75 | 77
SD | -0.1 (0.3) | 0 (0.2)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 16, analysis 1]; p = 0.11, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.1 to 0.0]

18. Secondary Outcome: Change in Waist Circumference
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 75 | 77
cm | 2.5 (7.7) | 2.3 (7.5)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Adjusted difference in mean changes in waist circumference (cm). The change in waist circumference is adjusted for the baseline waist circumference value; therefore, the adjusted difference in mean changes is not equal to the net change; Test type: Superiority — P-values and differences in mean changes from baseline were calculated using ANCOVA models, regressing changes from baseline to 52 weeks in waist circumference on treatment group and baseline value of waist circumference; p = 0.89, ANCOVA; Adjusted for baseline waist circumference (cm); Adjusted difference in mean changes = 0.2, 95% CI 2-sided [-2.3 to 2.6]

19. Secondary Outcome: Change in Fasting Serum Glucose
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 75 | 77
mg/dL | 1 (12) | 5 (27)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Adjusted difference in mean changes in fasting serum glucose. The change in fasting serum glucose is adjusted for the baseline fasting serum glucose value; therefore, the adjusted difference in mean changes is not equal to the net change; Test type: Non-Inferiority or Equivalence — P-values and differences in mean changes from baseline were calculated using ANCOVA models, regressing changes from baseline to 52 weeks in fasting serum glucose on treatment group and baseline fasting serum glucose value; p = 0.24, ANCOVA; Adjusted for baseline serum glucose value; Adjusted difference in mean changes = -4, 95% CI 2-sided [-11 to 3]

20. Secondary Outcome: Change in Fasting Insulin
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: μU/mL
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 75 | 77
μU/mL | 6 (36) | 10 (40)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Adjusted difference in mean changes in fasting insulin. The change in fasting insulin is adjusted for the baseline fasting insulin value; therefore, the adjusted difference in mean changes is not equal to the net change; Test type: Superiority — P-value and difference in mean changes from baseline were calculated using ANCOVA models, regressing changes from baseline to 52 weeks in fasting insulin on treatment group and baseline fasting insulin; p = 0.34, ANCOVA; Adjusted for baseline fasting insulin; Adjusted difference in mean changes = -6, 95% CI 2-sided [-18 to 6]

21. Secondary Outcome: Change in HOMA-IR
Description: (Glucose (mmol/L) x insulin (pmol/L))/22.5
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: (10E-15 mol^2)/L^2
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 75 | 77
(10E-15 mol^2)/L^2 | 1.4 (9.2) | 3.6 (12.5)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Adjusted difference in mean changes in HOMA-IR. The change in HOMA-IR is adjusted for the baseline HOMA-IR value; therefore, the adjusted difference in mean changes is not equal to the net change; Test type: Superiority — P-values and differences in mean changes from baseline were calculated using ANCOVA models, regressing changes from baseline to 52 weeks in HOMA-IR on treatment group and baseline HOMA-IR value; p = 0.15, ANCOVA; Adjusted for baseline HOMA-IR; Adjusted difference in mean changes = -2.6, 95% CI 2-sided [-6.2 to 1.0]

22. Secondary Outcome: Change in Systolic Blood Pressure
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 75 | 77
mmHg | 3 (12) | 2 (12)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Adjusted difference in mean changes in systolic blood pressure. The change in systolic blood pressure is adjusted for the baseline systolic blood pressure value; therefore, the adjusted difference in mean changes is not equal to the net change; Test type: Superiority — P-values and differences in mean changes from baseline were calculated using ANCOVA models, regressing changes from baseline to 52 weeks in systolic blood pressure on treatment group and baseline systolic blood pressure value; p = 0.71, ANCOVA; Adjusted for baseline systolic blood pressure; Adjusted difference in mean changes = 1, 95% CI 2-sided [-3 to 4]

23. Secondary Outcome: Change in Diastolic Blood Pressure
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 75 | 77
mmHg | -1 (9) | 1 (9)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Adjusted difference in mean changes in diastolic blood pressure. The change in diastolic blood pressure is adjusted for the baseline diastolic blood pressure value; therefore, the adjusted difference in mean changes is not equal to the net change; Test type: Superiority — P-values and differences in mean changes from baseline were calculated using ANCOVA models, regressing changes from baseline to 52 weeks in diastolic blood pressure on treatment group and baseline diastolic blood pressure value; p = 0.31, ANCOVA; Adjusted for baseline diastolic blood pressure; Adjusted difference in mean changes = -1, 95% CI 2-sided [-4 to 1]

24. Secondary Outcome: Change in Pediatric Quality of Life Inventory (PedsQL) Score
Description: Pediatric Quality of Life Inventory (PedsQL) version 4.0 is completed by both the child and parent/caregiver, and is composed of 23 items comprising 4 dimensions: Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning. Scores are transformed on a scale from 0 to 100, with higher scores indicating better health-related quality of life. Physical Health Summary Score =Physical Functioning Scale Score. Psychosocial Health Summary Score = Sum of items over the number of items answered in the Emotional, Social, and School Functioning Scales.
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 75 | 77
units on a scale
  Self-reported physical health | 4 (17) | 5 (16)
  Self-reported psychosocial health | 4 (15) | 5 (14)
  Parent/guardian-reported physical health | 4 (27) | 5 (24)
  Parent/guardian-reported psychosocial health | 5 (18) | 6 (24)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Adjusted difference in mean changes from baseline in self-reported Physical Health summary score from the Pediatric Quality of Life Inventory (PedsQL). The difference in mean changes in Physical Health summary score is adjusted for the baseline Physical Health summary score; therefore, the adjusted difference in mean changes is not equal to the net change. Higher scores indicate better health-related quality of life; Test type: Superiority — P-value and difference in mean changes from baseline were calculated using ANCOVA models, regressing changes from baseline to 52 weeks in self-reported Physical Health summary score on treatment group and baseline value of the Physical Health summary score; p = 0.77, ANCOVA; Adjusted for baseline self-reported Physical Health summary score; Adjusted difference in mean changes = -1, 95% CI 2-sided [-5 to 3]
Statistical Analysis 2: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Adjusted difference in mean changes from baseline in self-reported Psychosocial Health summary score from the Pediatric Quality of Life Inventory (PedsQL). The difference in mean changes in Psychosocial Health summary score is adjusted for the baseline Psychosocial Health summary score; therefore, the adjusted difference in mean changes is not equal to the net change. Higher scores indicate better health-related quality of life; Test type: Superiority — P-value and difference in mean changes from baseline were calculated using ANCOVA models, regressing changes from baseline to 52 weeks in Pyschosocial Health summary score on treatment group and baseline Psychosocial Health summary score; p = 0.64, ANCOVA; Adjusted for baseline Psychosocial Health summary score; Adjusted difference in mean changes = -1, 95% CI 2-sided [-5 to 3]
Statistical Analysis 3: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Adjusted difference in mean changes from baseline in parent/guardian-reported Physical Health summary score from the Pediatric Quality of Life Inventory (PedsQL). The difference in mean changes in parent/guardian-reported Physical Health summary score is adjusted for the baseline parent/guardian-reported Physical Health summary score; therefore, the adjusted difference in mean changes is not equal to the net change. Higher scores indicate better health-related quality of life; Test type: Superiority — P-value and difference in mean changes from baseline were calculated using ANCOVA models, regressing changes from baseline to 52 weeks in parent/guardian-reported Physical Health summary score on treatment group and baseline value of the parent/guardian-reported Physical Health summary score; p = 0.58, ANCOVA; Adjusted for baseline parent/guardian-reported Physical Health summary score; Adjusted difference in mean changes = -2, 95% CI 2-sided [-9 to 5]
Statistical Analysis 4: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Adjusted difference in mean changes from baseline in parent/guardian-reported Psychosocial Health summary score from the Pediatric Quality of Life Inventory (PedsQL). The difference in mean changes in parent/guardian-reported Psychosocial Health summary score is adjusted for the baseline parent/guardian-reported Psychosocial Health summary score; therefore, the adjusted difference in mean changes is not equal to the net change. Higher scores indicate better health-related quality of life; Test type: Superiority — P-value and difference in mean changes from baseline were calculated using ANCOVA models, regressing changes from baseline to 52 weeks in parent/guardian-reported Psychosocial Health summary score on treatment group and baseline value of the parent/guardian-reported Psychosocial Health summary score; p = 0.85, ANCOVA; Adjusted difference in mean changes = -1, 95% CI 2-sided [-6 to 5]

25. Secondary Outcome: Reduction in MRI-determined Hepatic Fat Fraction
Description: Change from baseline in MRI Proton Density Fat Fraction (PDFF) (%).
Time Frame: 52 weeks
Population: The smaller number of observations is because MRI was an optional procedure. This is the number with MRI exams at both baseline and 52 weeks.
Measure: Mean (Standard Deviation); unit: percentage of PDFF
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
Number analyzed (Participants) | 38 | 46
percentage of PDFF | -5.3 (7.1) | -2.6 (7.6)
Statistical Analysis 1: Comparison: DR Cysteamine Bitartrate Capsule vs DR Cysteamine Bitartrate Placebo; Test type: Superiority; p = 0.11, ANCOVA; Mean Difference (Final Values) = -2.7

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | DR Cysteamine Bitartrate Capsule | DR Cysteamine Bitartrate Placebo
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/81
Serious Adverse Events (participants affected / at risk) | 5/88 | 4/81
Other Adverse Events (participants affected / at risk) | 62/88 | 55/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DR Cysteamine Bitartrate Capsule (N=88) | DR Cysteamine Bitartrate Placebo (N=81)
Pain - Gallbladder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Infection - Appendix (Infections and infestations) | 0 (0) | 1 (1)
Mood alteration - depression (Psychiatric disorders) | 1 (2) | 1 (1)
Diabetes (Endocrine disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Personality/behavioral (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DR Cysteamine Bitartrate Capsule (N=88) | DR Cysteamine Bitartrate Placebo (N=81)
Pain - abdomen NOS (Gastrointestinal disorders) | 11 (11) | 8 (9)
Ocular - other (Eye disorders) | 1 (1) | 0 (0) — Change in prescription
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
Rhinitis (Immune system disorders) | 3 (3) | 5 (5)
Allergy - other (Immune system disorders) | 0 (0) | 1 (1) — Cat allergy
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mood alteration - anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 8 (10)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Teeth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diabetes (Endocrine disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 12 (12) | 11 (13)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pain - head/headache (Nervous system disorders) | 9 (9) | 6 (6)
Vomiting (Gastrointestinal disorders) | 6 (7) | 9 (10)
Pain - stomach (Gastrointestinal disorders) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (6)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (2)
Striae (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Infection - skin (Infections and infestations) | 1 (1) | 2 (2)
Pain - testicle (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Infection - urinary tract NOS (Infections and infestations) | 1 (1) | 1 (1)
Mood alteration - not specified (Psychiatric disorders) | 0 (0) | 2 (2)
Mood alteration - depression (Psychiatric disorders) | 2 (2) | 1 (1)
Mood alteration - irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Infection - ungual (Infections and infestations) | 2 (2) | 0 (0) — Nail infection
Hemorrhage - pulmonary - nose (General disorders) | 3 (5) | 4 (8) — Nosebleed
Pain - joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2)
Pain - breast (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metabolic/lab - other (Hepatobiliary disorders) | 0 (0) | 1 (1) — Increase in ALT and AST
Bone growth - spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hemorrhage, GI - rectum (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hemorrhage, GU - vaginal (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 3 (3)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 2 (2) | 3 (5)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Extremity - upper (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fever (Infections and infestations) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Metabolic/lab - other (Endocrine disorders) | 1 (1) | 0 (0) — Decrease in hemoglobin
Infection - pharynx (Infections and infestations) | 1 (1) | 1 (1)
Infection - larynx (Infections and infestations) | 0 (0) | 1 (1)
Infection - stomach (Infections and infestations) | 1 (1) | 1 (1)
Insomnia (General disorders) | 0 (0) | 1 (1)
Irregular menses (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Joint - function (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Lumbar spine ROM (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal/paranasal reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infection - middle ear (otitis media) (Infections and infestations) | 4 (5) | 3 (3)
Pain - middle ear (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Pain - skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain - chest wall (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain (extremity - limb) (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4)
Pain - bone (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Ocular surface disease (Eye disorders) | 0 (0) | 1 (1)
Ocular - other (Eye disorders) | 0 (0) | 1 (1) — Periorbital cellulitis
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Infection (middle ear) with unknown ANC (Infections and infestations) | 1 (1) | 0 (0)
Infection (ungual) with unknown ANC (Infections and infestations) | 0 (0) | 1 (1)
Infection (sinus) with unknown ANC (Infections and infestations) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Infection - upper airway NOS (Infections and infestations) | 3 (4) | 3 (3)
Sexual - other (orchiopexy) (Surgical and medical procedures) | 0 (0) | 1 (1)
Pulmonary - other (cold) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Infection - bronchus (Infections and infestations) | 0 (0) | 1 (1)
Dermatology - other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Edematous nodular lesions with pruritus
Flu-like syndrome (General disorders) | 3 (3) | 0 (0)
Dermatology - other (warts, HPV) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Infection - sinus (Infections and infestations) | 0 (0) | 1 (1)
Infection (documented clinically) - pharynx (Infections and infestations) | 1 (1) | 0 (0)
Infection - lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pulmonary - other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Positive PPD, negative chest X-ray
Metabolic/lab - other (Endocrine disorders) | 1 (1) | 0 (0) — Worsening insulin resistance
Neuropathy - sensory (Nervous system disorders) | 2 (2) | 0 (0)
Neurology - other (concussion) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint - function (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Intraop injury - liver (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pain - throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dermatology - other (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Stepped on nail
Musculoskeletal - other (ankle sprain) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Musculoskeletal - other (wrist sprain) (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Musculoskeletal - other (finger sprain) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical spine ROM (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Musculoskletal - other (spondylosis) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 2 (2)
Ocular - other (eye redness, allergies) (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No